CLINICAL TRIAL: NCT04321434
Title: Cardiac and Subcutaneous Microvascular Dysfunction in Patients With Ischemic Heart Disease: Effects of an Acute Oxidative Stress
Brief Title: Hyperoxia and Microvascular Dysfunction
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Futility
Sponsor: Université Libre de Bruxelles (Other)
Responsible Party: Principal Investigator, Martin Chaumont, Principal investigator, Université Libre de Bruxelles
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: P2016/043/B406201627021
Record Dates: First submitted 2017-01-16; First posted 2020-03-25 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Coronary Microvascular Disease; Microvascular Disease; Ischemic Heart Disease
Keywords: cardiac microvascular dysfunction; subcutaneous microvascular dysfunction; ischemic heart disease; oxydative stress
MeSH Terms: conditions — Microvascular Angina; Myocardial Ischemia | interventions — Laser-Doppler Flowmetry

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hyperoxia (Experimental): * assessment of forearm skin microcirculatory blood flow by laser Doppler perfusion imager at baseline and during hyperemic tests
  * assessment of coronary microcirculatory blood flow at baseline and during hyperemic tests
  Interventions: Other: Hyperoxia; Device: laser Doppler
- Normoxia (Placebo Comparator): * assessment of forearm skin microcirculatory blood flow by laser Doppler perfusion imager at baseline and during hyperemic tests
  * assessment of coronary microcirculatory blood flow at baseline and during hyperemic tests
  Interventions: Other: Normoxia; Device: laser Doppler

INTERVENTIONS:
Other: Hyperoxia
  Arms: Hyperoxia
Other: Normoxia
  Arms: Normoxia
Device: laser Doppler — laser Doppler

SUMMARY:
Coronary artery disease (CAD) pathophysiology involves endothelium-dependent (e.g. nitric oxide, acetylcholine) and -independent (e.g. adenosine) vascular dilation impairment, which have been demonstrated at the level of small coronary arteries, medium sized peripheral arteries and subcutaneous microcirculation. Oxygen supplementation, which is frequently overused in clinical settings, seems harmful in acute coronary syndromes and increases microvascular resistance in myocardial and subcutaneous microcirculation through alteration of endothelium-dependent and -independent dilation by an oxidative mechanism. Whether endothelial dysfunction, that is well documented at the level of cardiac microcirculation in CAD patients, is also present at the level of subcutaneous microcirculation is unknown. Also, unknown is whether an acute oxidative stress can be used to probe myocardial microcirculatory dysfunction at the level of subcutaneous microcirculation, which is an easily accessible vascular bed for an in vivo assessment of endothelial-dependent and-independent function. Alterations in cutaneous vascular signalling are evident early in the disease processes. Thus, studying subcutaneous circulation in patients with cardiovascular risk factors could provide vascular information early in CAD processes. This study will test the following 4 hypotheses:

1. Endothelial dysfunction observed at the level of microvascular cardiac arteries is readily present at the level of subcutaneous microcirculation in a given CAD patient.
2. An acute oxidative stress such as hyperoxia can be used to test myocardial microcirculatory dysfunction at the level of the more easily accessible subcutaneous microcirculation.
3. Subcutaneous microcirculation of CAD patients has a lesser vasodilatory response to acetylcholine or sodium nipride than matched healthy subjects. In addition, CAD patients are more prone to dermal vasoconstriction in response to oxygen compared to healthy subjects.
4. Taken that oxygen is still too often given in excess in most clinical settings, the aim of this study is to rule out possible pitfalls in coronary pressure and resistance determinations in CAD patients receiving unnecessary oxygen supplementation.

ELIGIBILITY:
Inclusion Criteria:

* Coronary angiography done in the context of suspicion of coronary artery disease (CAD)

Exclusion Criteria:

* Respiratory failure requiring intubation or supplementary oxygen
* Severe chronic obstructive pulmonary disease
* Significant arrhythmia precluding waveform analysis (e.g., excessive premature ventricular contractions or atrial fibrillation)
* Severe valvular heart disease,
* Suspected elevated central venous pressure (CVP)
* Heart failure as defined by New York Heart Association class III or IV
* Previous coronary revascularization or heart transplantation
* Severe hypertension (systolic pressure >200 mmHg and diastolic pressure >120 mmHg at rest)
* Contraindications to adenosine infusion
* Contraindication to acetylcholine (Ach) infusion
* Severe bronchial asthma.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-12-01; Primary Completion 2018-04-01 (Actual); Study Completion 2018-10-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the acetylcholine-induced skin blood flow after hyperoxia | 1 hour
  Measurement of skin blood flow before, during and after hyperoxia, expressed in perfusion units (arbitrary units).
Change from baseline in the sodium nitroprusside-induced skin blood flow after hyperoxia | 1 hour
  Measurement of skin blood flow before, during and after hyperoxia, expressed in perfusion units (arbitrary units).
Change from baseline in the heat-induced skin blood flow after hyperoxia | 1 hour
  Measurement of skin blood flow before, during and after hyperoxia, expressed in perfusion units (arbitrary units).
Change from Baseline in the index of microcirculatory resistance Under adenosine after hyperoxia | 10 minutes
  Measurement of coronary microcirculatory resistance (index of microcirculatory resistance) Under adenosine before and after hyperoxia, expressed in arbitrary units
Change from Baseline in the index of microcirculatory resistance at rest after hyperoxia | 10 minutes
  Measurement of coronary microcirculatory resistance (index of microcirculatory resistance) at rest before and after hyperoxia, expressed in arbitrary units

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Paul Van Vooren, MD, PhD, Study Director — Hospital Erasme
Locations (1):
- Erasme Hospital, Brussels, Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No